CLINICAL TRIAL: NCT06917469
Title: Use of New MolEcular MarkErs for a persoNalized Therapy in Ovarian Cancer-MEMENTO
Acronym: MEMENTO
Status: Completed | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2018-38
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ovarian cancer (OC) is the leading cause of death from gynecologic cancer. It is estimated that 22,440 new cases of EOC will be diagnosed in 2017 with an estimated 14,080 EOC deaths. Several different histological subtypes of OC can be identified.

Over 90% of malignant ovarian tumors are epithelial cancers (EOC), which are then classified into 5 broad histological subtypes: serous, endometrioid, mucinous, clear cell and mixed or carcinosarcomatous mullerian tumors. Almost 10 years ago, a new classification was proposed that separated ovarian cancers into type I and II tumors.

Type II tumors included high-grade serous, which frequently contain mutations in p53, NF1, BRCA1, and BRCA2 and CDK125. Serous carcinomas represent the vast majority of primary malignant ovarian tumors (75%-80%), among these high-grade serous (HGSOC) accounts for 85%-90% and for the majority of the deaths due to ovarian cancer. The 5-year survival rate for EOC is only 46% because >60% of patients are diagnosed with advanced disease. Patients with advanced stage EOC are typically managed with cytoreductive surgery and perioperative platinum-based chemotherapy, either in the adjuvant setting or with neoadjuvant chemotherapy and interval debulking surgery.

Although primary advanced stage EOC is initially sensitive to this treatment paradigm, >75% will eventually recur. Patients with recurrent disease are treated with additional lines of chemotherapy that may increase survival but is ultimately not curative. Given the high relapse rate and poor prognosis of advanced stage EOC, interest is increasing in the development of new approaches to treat recurrent EOC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of a first relapse of high-grade ovarian cancer (≥12 months after the last platinum administration);
* p53 positive tumors evaluated by IHC (>30% of stained tumor cells);
* Performance Status (Eastern Cooperative Oncology Group scale, ECOG) ≤ 2;- Availability of the tumor sample for immunohistochemical analysis;
* Written informed consent.

Exclusion Criteria:

* Pre-existing or concurrent tumors, except in situ carcinoma or basophilic carcinoma of the skin;
* Low p53 expression levels (<30% of stained tumor cells);
* Persistent grade≥ 2 neuropathy;
* Severe heart disease;
* Surgeon's decision of a second curative surgery;
* Uncontrolled active infections;
* Insufficient patient compliance;
* Absence of signed informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with histological diagnosis of high-grade ovarian carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
To assess DNA-PK as a potential predictive biomarker for distinguishing patients who will benefit from CBDCA/TAX therapy from those who will respond more favorably to the CBDCA/PLD regimen, based on DNA-PK expression levels. | up to 5 years
  Two years progression free survival will be estimated with Kaplan-Meier methods and reported as survival probability in the two treatment groups. PFS will be defined as time from the beginning of second line platinum based therapy and progression or death or end of follow-up whichever comes first

SECONDARY OUTCOMES:
Evaluation of the Response Rate | up to 5 years
  Response rate will be reported as numbers and percentages and evaluated based on RECIST 1.1 criteria
Evaluation of Overall Survival in the different treatment regimens | Up to 5 years
  Overall Survival (OS) will be evaluated with Kaplan-Meier methods and reported separately for the two treatment groups. OS will be defined as time from the beginning of second line platinum based therapy and death or end of follow-up whichever comes first
PFS in patients treated with biomarker driven therapy and physician's choice therapy | up to 5 years
  Difference in PFS between subgroups of patients will be evaluated with Kaplan-Meier method and log-rank test
OS in patients treated with biomarker driven therapy and physician's choice therapy | up to 5 years
  Difference in OS between subgroups of patients will be evaluated with Kaplan-Meier method and log-rank test

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Riferimento Oncologico - IRCCS, Aviano, Italy